CLINICAL TRIAL: NCT06104345
Title: Immune Response Elicited by Concomitant Administration of Oral Typhoid Fever (Vivotif®) and Cholera (Dukoral®) Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Anu Kantele, MD, PhD, Professor of Infectious Diseases, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dukoral+Vivotif
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Vaccine-Preventable Diseases; Typhoid Fever; Cholera
Keywords: Immunogenicity; Coadministration; ELISPOT; B cells; Oral vaccination; Salmonella Typhi; Vibrio cholerae
MeSH Terms: conditions — Vaccine-Preventable Diseases; Typhoid Fever; Cholera | interventions — Ty21a typhoid vaccine; Cholera Vaccines; Dukoral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vivotif (Active Comparator): Three oral doses of typhoid fever vaccine (Vivotif®).
  Interventions: Biological: Oral typhoid fever vaccine
- Dukoral (Active Comparator): Two oral doses of cholera vaccine (Dukoral®).
  Interventions: Biological: Oral cholera vaccine
- Dukoral+Vivotif (Experimental): Oral typhoid fever and cholera vaccines (Vivotif® and Dukoral®) administered simultaneously.
  Interventions: Biological: Oral typhoid fever vaccine; Biological: Oral cholera vaccine

INTERVENTIONS:
Biological: Oral typhoid fever vaccine — Oral typhoid fever vaccine (Vivotif®) on Days 0, 2 and 4.
  Other Names: Vivotif®
  Arms: Dukoral+Vivotif; Vivotif
Biological: Oral cholera vaccine — Oral cholera vaccine (Dukoral®) on Days 0 and 7.
  Other Names: Dukoral®
  Arms: Dukoral; Dukoral+Vivotif

SUMMARY:
The goal of this clinical trial is to explore the coadministration of oral typhoid fever (Vivotif®) and cholera (Dukoral®) vaccines in healthy volunteers aged 18-65 years. The main question it aims to answer is:

• Does coadministration impact the immune responses to Vivotif® and Dukoral® vaccines

Participants will:

* receive either oral typhoid fever (Vivotif®) or oral cholera (Dukoral®) vaccines or both simultaneously
* give blood samples for immunogenicity analyses
* participate in adverse event follow up

Researchers will compare those receiving only one of the vaccines to those receiving both simultaneously to see if coadministration has an impact on antigen-specific responses measured with:

* ELISPOT (plasmablast responses specific to Salmonella typhi, Vibrio Cholerae and Enterotoxigenic Escherichia coli)
* ELISA (antibodies in lymphocyte supernatants (ALS) and serum antibodies specific to vaccine antigens)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 to ≤65 years.
2. General good health as established by medical history and physical examination.
3. Written informed consent.
4. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study (14 days before immunization to day 28 ± 3). Abstinence is acceptable.
5. Available for all visits scheduled in this study.

Exclusion Criteria:

1. Vaccination against typhoid fever or cholera within 5 years before dosing.
2. History of clinical typhoid fever or cholera.
3. Immunization with any other vaccine (oral or parenteral) within 4 weeks prior to study period or vaccination planned during it.
4. Current intake of antibiotics or end of antibiotic therapy <8 days before first IMP administration.
5. Chronic (longer than 14 days) administration of immunosuppressants or other immunemodifying drugs within 6 months before the first dose of IMP; oral corticosteroids in dosages of ≥0.5 mg/kg/d prednisolone or equivalent are excluded; inhaled or topical steroids allowed.
6. Acute or chronic clinically significant gastrointestinal disease.
7. Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
8. Pregnancy or lactation.
9. Acute disease at the time of enrolment (defined as the presence of a moderate or severe illness with or without fever (fever defined as body temperature of ≥38 °C).
10. Alcohol or drug abuse.
11. Suspected non-compliance.
12. Use of any investigational drug or vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
13. Any clinically significant history of known or suspected anaphylaxis or hypersensitivity reaction based on the judgement of the investigator.
14. Employee at the investigational site or relative or spouse of the investigator.
15. Any other criteria which, in the investigator's opinion, would compromise the ability of a subject to participate in the study, a subject's well-being, or the outcome of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Magnitude of antigen-specific plasmablast responses to oral typhoid fever (Vivotif®) and cholera (Dukoral®) vaccines (ASCs/million PBMCs) | Blood samples on Days 0-7 for all participants and Days 12-14 for participants in Dukoral and Dukoral+Vivotif arms.
  Measurement of IgA -, IgG- and IgM-secreting antibody cells (ASC ELISPOT) specific to Salmonella typhi (whole cell), Vibrio cholerae (whole cell and CTB-toxin) and Enterotoxigenic Escherichia coli (ETEC whole cell and LTB-toxin).

SECONDARY OUTCOMES:
Titer of antigen-specific antibodies in lymphocyte supernatants (ALS) to oral typhoid fever (Vivotif®) and cholera (Dukoral®) vaccines. | Blood samples on Days 0-7 for all participants and Days 12-14 for participants in Dukoral and Dukoral+Vivotif arms.
  Measurement of anti-salmonella, anti-cholera and anti-ETEC antibodies in ALS samples (ELISA)

OTHER OUTCOMES:
Titer of antigen-specific serum antibodies to oral typhoid fever (Vivotif®) and cholera (Dukoral®) vaccines. | Blood samples on Days 0 and 28 ± 3 for all participants.
  Measurement of anti-salmonella, anti-cholera and anti-ETEC antibodies in serum (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Anu Kantele, MD, PhD, Principal Investigator — Meilahti Vaccine Research Center, MeVac, Helsinki University Hospital
Locations (1):
- Meilahti Vaccine Research Center, Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
The decision to share IPD will be done when the study is completed. IPD can be shared only if it does not compromise the anonymity of the study participants.